CLINICAL TRIAL: NCT07019194
Title: An Open-label, Randomized, Single-dose, Two-way Crossover Bioequivalence Study to Compare Two Strengths (10 mg and 20 mg) of Senaparib Capsules in Healthy Chinese Subjects Following Oral Administration Under Fasting Condition
Brief Title: An Bioequivalence Study to Compare 10mg & 20mg of Senaparib Capsules in Healthy Chinese Subjects Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IMP4297-113
Record Dates: First submitted 2025-05-23; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor
MeSH Terms: interventions — senaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Senaparib capsules first 1*20mg then 2*10mg (Experimental): Single oral dose of Senaparib administered under fasting condition, 1*20mg capsules in first intervention period and then 2*10mg capsules in second intervention period (after washout period: at least 5 days)
  Interventions: Drug: Senaparib capsules(20mg); Drug: Senaparib capsules(10mg)
- Senaparib capsules first 2*10mg then 1*20mg (Experimental): Single oral dose of Senaparib administered under fasting condition, 2*10mg capsules in first intervention period and then 1*20mg capsules in second intervention period (after washout period: at least 5 days)
  Interventions: Drug: Senaparib capsules(20mg); Drug: Senaparib capsules(10mg)

INTERVENTIONS:
Drug: Senaparib capsules(20mg) — Single oral dose of Senaparib administered under fasting condition, 1*20mg capsules in first intervention period and then 2*10mg capsules in second intervention period (after washout period: at least 5 days)
Drug: Senaparib capsules(10mg) — Single oral dose of Senaparib administered under fasting condition, 2*10mg capsules in first intervention period and then 1*20mg capsules in second intervention period (after washout period: at least 5 days)

SUMMARY:
An Open-label, Randomized, Single-dose, Two-way Crossover Bioequivalence Study to Compare Two Strengths (10 mg and 20 mg) of Senaparib Capsules in Healthy Chinese Subjects Following Oral Administration Under Fasting Condition

DETAILED DESCRIPTION:
An Open-label, Randomized, Single-dose, Two-way Crossover Bioequivalence Study to Compare Two Strengths (10 mg and 20 mg) of Senaparib Capsules in Healthy Chinese Subjects Following Oral Administration Under Fasting Condition.

It was planned to enroll 40 subjects in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understood the purpose, nature, methods and possible adverse reactions of the trial, voluntarily participated in the trial, and signed an informed consent form (ICF) before any trial procedure, and promised to participate in all procedure of the trial.
2. Healthy Chinese male subjects aged 18 to 55 (inclusive) at screening.
3. Body mass index (BMI) ranged from 19.0 to 27.0 kg/m2 (inclusive); body weight ≥ 50.0 kg.
4. Vital signs measurement [reference range (inclusive): systolic blood pressure 90 to 140 mmHg, diastolic blood pressure 60 to 90 mmHg, pulse 50 to 100 bpm, body temperature (ear temperature) 35.8 to 37.2°C], comprehensive physical examination, other clinical laboratory tests during the screening period and auxiliary examination showed normal or abnormal results by the investigator without clinical significance.
5. Subjects could communicate well with the investigators and understood and abided by the requirements of this trial.

Exclusion Criteria:

1. (Inquiry) Subjects with diseases with clinical abnormality, including but not limited to disease concerning nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolic system and skeletal system.
2. (Inquiry) Subjects with allergic history (including drug and food allergies, etc.) and allergy to Senaparib capsules or any component of the drug product.
3. (Inquiry) Subjects with history of dysphagia or any gastrointestinal disease that affected drug absorption judged by the investigator.
4. (Inquiry) Subjects who had received surgery within 3 months before screening, or planned to have surgery during the trial period, or those who had previous surgery that would affect drug absorption (e.g. gastrectomy).
5. (Inquiry) Subjects who could not tolerate venipuncture, or had a history of needlesickness and fainting at the sight of blood.
6. (Inquiry) Subjects who had drug abuse history within 6 months before screening.
7. (Inquiry) Subjects who consumed more than 14 units of alcohol per week (1 unit of alcohol = 360 mL beer, 150 mL wine, or 45 mL liquor) within 3 months before screening, or could not give up alcohol during the trial.
8. (Inquiry) Subjects who consumed an average of more than 5 cigarettes per day within3 months before screening, or who could not stop using any tobacco products during the trial.
9. (Inquiry) Subjects who consumed an average of excessive amounts of tea, coffee and/ or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) every day within 3 months before screening.
10. (Inquiry) Subjects who had participated in clinical trials of other study drugs/devices within 3 months before screening (if other study drugs had a longer half-life, the time interval would be longer and was required to be 5 half-lives of the drug), or had participated in 3 or more clinical trials of drugs/devices in the past year.
11. (Inquiry) Subjects who donated blood including blood component or had massive blood loss (≥ 400 mL), or received blood transfusion or used blood products and blood biological products within 3 months before screening.
12. (Inquiry) Subjects who received live vaccines within 4 weeks before screening.
13. (Inquiry) Subjects who had taken any drugs [such as: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; SSRI(selective serotonin reuptake inhibitor) antidepressants, cimetidine, macrolides, nitroimidazoles, sedative hypnotics, fluoroquinolones, antihistamines, antivirals (such as saquinavir), calcium antagonists (such as diltiazem, verapamil), rifamycins (such as rifampicin)] that inhibit or induce the liver to metabolize drug within 28 days before screening. If the past drug used had a longer half-life, the time interval would be longer and was required to be 5 half-lives of the drug, e.g., phenobarbital required a 5-week washout period.
14. (Inquiry) Subjects who had taken prescription drugs, over-the-counter drugs, dietary supplements or Chinese herbal medicine within 14 days before screening. If the past drug used had a longer half-life, the time interval would be longer and was required to be 5 half-lives of the drug.
15. At screening, the corrected QT interval (corrected by Fridericia's formula, QTcF(Corrected QT interval using Fridericia's fomula) = QT/RR1/3) > 450 msec or QRS complex > 120 msec was obtained by 12-lead ECG in supine position in resting state, or the presence of other clinically significant abnormalities was judged by the investigator.
16. (Inquiry) Vigorous exercise could not be avoided within 48 hours before the first dose of the investigational drug and during the trial.
17. (Inquiry) Subjects who could not abstain from any food or beverages containing alcohol, caffeine, chocolate, or rich in xanthine within 48 hours before the first dose of the investigational drug and during the trial.
18. (Inquiry) Subjects who could not abstain from grapefruit or grapefruit-related citrus (e.g., pomelo) or juice within 7 days before the first dose of investigational drug and during the trial.
19. (Inquiry) Subjects or its partners who had birth plan, or were unwilling to adopt effective contraception methods, or had sperm donation plan throughout the trial and within 90 days after the last dose of the investigational drug.
20. (Inquiry) Subjects who were unwilling or unable to follow the lifestyle guidelines described in the study protocol (such as dietary restrictions and activity requirements).
21. Subjects judged by the investigator to be unsuitable for participation in the trial.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-48 hour
  Maximum concentration.
AUC0-last | 0-48 hour
  area under the curve from time 0 to the last time with quantifiable concentration
AUC0-inf | 0-48 hour
  if the data were available, area under the curve from time 0 to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Chaolin Huang, Principal Investigator — Wuhan Jinyintan Hospital (Wuhan Infectious Disease Hospital)
Locations (1):
- Wuhan Jinyintan Hospital (Wuhan Infectious Disease Hospital), Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No